CLINICAL TRIAL: NCT04762459
Title: Efficacy and Safety of Almonertinib Combined With or Without Chemotherapy as an Adjuvant Treatment for EGFR Mutation Positive Stage II-IIIA Non-small Cell Lung Carcinoma Following Complete Tumour Resection: A Multicenter, Randomized Controlled, Open-label Clinical Study
Brief Title: Efficacy and Safety of Almonertinib Combined With or Without Chemotherapy as an Adjuvant Treatment for Stage II-IIIA Non-small Cell Lung Carcinoma Following Complete Tumour Resection
Acronym: APEX
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry); GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shugeng Gao, Chief Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YX-L-202105
Record Dates: First submitted 2021-02-10; First posted 2021-02-21 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2021-02

CONDITIONS: Non-small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Almonertinib (Active Comparator): Drug: Almonertinib 110 mg A cycle of treatment is defined as 21 days of once daily treatment. Number of Cycles: The patient continues to receive treatment until the disease progresses or reaches termination criteria. The overall treatment last for 3 years.
  Interventions: Drug: Almonertinib
- Almonertinib/Pemetrexed/Cisplatin (Experimental): Drug: Almonertinib 110 mg Drug: Pemetrexed 500 mg/m² IV on day 1 of each 21 day cycle. Number of cycles until disease progression or unacceptable toxicity develops.
  Drug: Cisplatin 75mg/m2 IV on day 1 of each 21 day cycle. Number of cycles until disease progression or unacceptable toxicity develops.
  A cycle of treatment is defined as 21 days of once daily treatment. Number of Cycles: The patient continues to receive treatment until the disease progresses or reaches termination criteria. The overall treatment last for 3 years.
  Interventions: Drug: Almonertinib; Drug: Pemetrexed; Drug: Cisplatin
- Pemetrexed/Cisplatin (Active Comparator): Drug: Pemetrexed 500 mg/m² IV on day 1 of each 21 day cycle. Number of cycles until disease progression or unacceptable toxicity develops.
  Drug: Cisplatin 75mg/m2 IV on day 1 of each 21 day cycle. Number of cycles until disease progression or unacceptable toxicity develops.
  A cycle of treatment is defined as 21 days of once daily treatment. Number of Cycles: The patient continues to receive treatment until the disease progresses or reaches termination criteria. If disease progresses during the treatment period and conditions required for the cross-treatment are met according to the assessment process, the patient can start to receive the open cross-treatment of Almonertinib. The overall treatment last for 3 years.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Almonertinib — Almonertinib 110mg PO once daily
  Arms: Almonertinib; Almonertinib/Pemetrexed/Cisplatin
Drug: Pemetrexed — 500 milligrams per square meter (mg/m²) Pemetrexed
  Arms: Almonertinib/Pemetrexed/Cisplatin; Pemetrexed/Cisplatin
Drug: Cisplatin — 75mg/m² Cisplatin taken intravenously (IV) once every 3 weeks concurrently
  Arms: Almonertinib/Pemetrexed/Cisplatin; Pemetrexed/Cisplatin

SUMMARY:
This is a multicenter, randomized, open label, phase III study.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open label, phase III study assessing the efficacy and safety of Almonertinib combined with or without chemotherapy as an adjuvant treatment in patients with epidermal growth factor receptor (EGFR) mutation positive stage II-IIIA non-squamous NSCLC following complete tumour resection: Eligible patients will be randomized to receive either Almonertinib alone (110mg, po, once daily) or Almonertinib (110mg, po, once daily) plus pemetrexed (500mg/m2, iv) and cisplatin (500mg/m2, iv) or pemetrexed (500mg/m2, iv) plus cisplatin (500mg/m2, iv) in a 3:2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who meets all of the following inclusion criteria will qualify for entry into the study:

  1. Male or female, aged at least 18 years.
  2. Histologically confirmed diagnosis of primary non small lung cancer (NSCLC) on predominantly non-squamous histology.
  3. Brain examination must be done prior to surgery as it is considered standard of care.
  4. Patients must be classified post-operatively as Stage II-IIIA on the basis of pathologic criteria.
  5. Confirmation by the central laboratory that the tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations including T790M.
  6. Providing paraffin embedded section(10-15sheets),wax blocks or fresh frozen tissues.
  7. Complete surgical resection of the primary NSCLC is mandatory. All gross disease must have been removed at the end of surgery. All surgical margins of resection must be negative for tumour.
  8. World Health Organization Performance Status of 0 to 1.
  9. Women of childbearing age should take appropriate contraceptive measures from screening to 3 months after stopping the study treatment and should not breastfeed. Before starting the administration, the pregnancy test was negative.
  10. Male patients should be willing to use barrier contraception from screening to stopping study treatment for 3 months.(i.e., condoms).
  11. For inclusion in study, patient must provide a written informed consent.
  12. ≤10 weeks between surgery and randomization.

Exclusion Criteria:

* Any patient who meets any of the following exclusion criteria will not qualify for entry into the study:

  1. Treatment with any of the following:

     1. Pre-operative or post-operative or planned radiation therapy for the current lung cancer
     2. Pre-operative (neo-adjuvant) platinum based or other chemotherapy
     3. Prior treatment with neoadjuvant or adjuvant EGFR-TKI at any time
     4. Any other anti-tumor treatment for lung cancer(Including proprietary Chinese patent medicine with anti-tumor effects and anti-tumor immunotherapy, etc.)
     5. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
     6. Treatment with an investigational drug within five half-lives of the compound or any of its related material.
     7. Medications that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug..
  2. Patients who have had only segmentectomies or wedge resections
  3. History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer, or other solid tumours curatively treated with no evidence of disease for > 5 years following the end of treatment.
  4. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
  5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
  6. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of Almonertinib.
  7. Any of the following cardiac criteria:

     1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
     2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
     3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
  8. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
  9. Inadequate bone marrow reserve or organ function.
  10. History of hypersensitivity to any active or inactive ingredient of Almonertinib, or to drugs with a similar chemical structure or class to Almonertinib.
  11. Patients who are allergic to pemetrexed or any other ingredients in the preparation, cisplatin or other platinum-containing compounds.
  12. Patients with contraindications of pemetrexed and cisplatin.
  13. Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.
  14. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
  15. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Defined as the time from the date of randomization until the date of disease recurrence or death (by any cause in the absence of recurrence)

SECONDARY OUTCOMES:
Disease free survival (DFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Defined as the proportion of patients alive and disease free at 2, 3 ,4and 5 years, respectively, estimated from Kaplan Meier plots of the primary endpoint of DFS at the time of the primary analysis.
Overall Survival (OS) | Start of study drug to Survival Endpoint through study completion, an average of 5 years, assessed up to 100 months
  Defined as the time from the date of randomization until date of death due to any cause.
Patient health-related quality of life and symptoms (HRQoL) by SF-36v2 Health Survey | From date of randomization until treatment completion or discontinuation, assessed up to 100 months
  Defined as a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section and the scores range from 0-100. A score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.

OTHER OUTCOMES:
Incidence of Adverse Events (AEs) | From date of randomization until 28 days after treatment completion
  AEs graded by CTCAE version 4.0

CONTACTS AND LOCATIONS:
Locations (34):
- China (34):
  - Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chendu
  - Sichuan Provincial People's Hospital, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Consonancy Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University School Of Medicine, Hangzhou
  - The First People's Hospital of Yunnan Province, Kunming
  - Yunnan Cancer Hospital, Kunming
  - JiangXi Cancer Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Provincial People's Hospital, Nanjing
  - Ningbo Medical Center Li Huili Hospital, Ningbo
  - Qingdao Municipal Hospital, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - ShangHai Chest Hospital ShangHai JiaoTong University, Shanghai
  - ShangHai Pulmonary Hospital, Shanghai
  - Liaoning Cancer Hospital, Shenyang
  - Cancer Hospital Chinese Academy of Medical Sciences,Shenzhen Center, Shenzhen
  - Hebei Cancer Hospital, Shijiazhuang
  - West China Hospital，Sichuan University, Sichuan
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Thoracic Surgery Department Of The ShanXi Provincial Cancer Hospital, Taiyuan
  - Tianjin Chest Hospital, Tianjin
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi
  - Weifang People's Hospital, Weifang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Union Hospital Of China, Wuhan
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou